CLINICAL TRIAL: NCT05350891
Title: A Prospective, Single-arm, Multicenter Clinical Study of Transnasal Endoscopic Surgery Combined With Adjuvant Immunotherapy for Recurrent Nasopharyngeal Carcinoma
Brief Title: Transnasal Endoscopic Surgery Combined With Adjuvant Immunotherapy for Recurrent NPC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Collaborators: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Hongmeng Yu, Principal Investigator, Professor, Eye & ENT Hospital of Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: rNPC-SA-Ad-Immuno-V1
Record Dates: First submitted 2022-03-22; First posted 2022-04-28 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Recurrent Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Endoscopy; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- endoscopic surgery combined with adjuvant immunotherapy (Experimental)
  Interventions: Procedure: endoscopic surgery

INTERVENTIONS:
Procedure: endoscopic surgery — endoscopic surgery combined with adjuvant immunotherapy with/without chemotherapy
  Other Names: adjuvant immunotherapy; chemotherapy

SUMMARY:
A Prospective, Single-arm, Multicenter Clinical Study of Transnasal Endoscopic Surgery Combined With Adjuvant Immunotherapy for Recurrent Nasopharyngeal Carcinoma

ELIGIBILITY:
Inclusion Criteria:

* Pathology or radiography confirmed recurrent nasopharyngeal carcinoma.
* AJCC rT1-T4 which can be surgically removed.
* Age ≥18 years old.
* Informed consent signed.
* With or without lymph node metastasis, which can be surgically removed.
* No distant metastasis.
* ≥6 months from the end of initial radiotherapy to recurrence.
* Sufficient organ function a)Hematology: white blood cells ≥3.0 x 109/L, absolute neutrophil count ≥1.5x 109/L, hemoglobin ≥80 g/L, platelets ≥100 x 109/L. b) Liver function: bilirubin ≤ 1.5 times the upper limit of normal (ULN), AST and ALT ≤ 3 times the ULN c) International normalized ratio (INR) or prothrombin time (PT) or activated partial thromboplastin time (aPTT) ≤ 1.5 times ULN. d) Renal function: serum creatinine ≤ 1.5 times ULN.
* ECOG score 0-2. general physical condition can tolerate general anesthesia surgery, chemotherapy, and immunotherapy.

Exclusion Criteria:

* Evidence of distant metastasis or leptomeningel disease (LMD).
* Have received radioactive seed implantation in the treatment area.
* Suffer from uncontrolled disease which could interfere with treatment.
* Suffered from another malignant tumor or multiple primary tumors at the same time within 5 years (excluding fully treated basal cell or squamous cell skin cancer, cervical cancer in situ, etc.).
* The patient has surgical contraindications: such as severe cardiopulmonary disease, coagulation dysfunction and so on.
* The patients have autoimmune diseases.
* The patient is using immunosuppressive agents or systemic glucocorticoid to achieve the purpose of immunosuppression (dose>10mg/day prednisone or other), and continues to use it within 2 weeks before the first administration.
* Severe allergic reaction to other monoclonal antibodies.
* Previously received PD-1 monoclonal antibody, CTLA-4 monoclonal antibody (or any other antibody that acts on T cell co-stimulation or checkpoint pathway) treatment.
* Live vaccines have been inoculated within 4 weeks before the first administration or during the study period.
* The patient has any situation that may hinder study compliance or the safety during the study period.
* Existence of serious neurological or psychiatric diseases, such as dementia and seizures.
* Uncontrolled active infection.
* Pregnant or breastfeeding women.
* Those who have no personal freedom and independent capacity for civil conduct.
* There are other situations that are not suitable for entry into the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Estimated)
Dates: Start 2022-05-08 (Estimated); Primary Completion 2026-05-08 (Estimated); Study Completion 2026-05-08 (Estimated)

PRIMARY OUTCOMES:
progression free survival | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first，through study completion,up to 2 years.
  2 year progression free survival

SECONDARY OUTCOMES:
Overall survival | From date of enrollment until the date of death from any cause,through study completion,up to 2 years.
  2 year Overall Survival rate

OTHER OUTCOMES:
Local progression free survival | From date of enrollment to local failure or date of death from any cause,through study completion,up to 2 years.
  2 year Local progression free survival
Distant metastasis free survival | From date of enrollment to distant metastasis or date of death from any cause, through study completion,up to 2 years.
  2 year distant metastasis free survival
Toxicities | From date of enrollment through study completion,up to 2 years.
  Using CTCAE Version5.0 to evaluate incidence of Treatment-Related Adverse Events including treatment related adverse effect and immune related adverse effect.

CONTACTS AND LOCATIONS:
Overall Officials: Hongmeng Yu, MD,PHD, Principal Investigator — Eye&ENT Hospital,Fudan University
Locations (8):
- China (8):
  - The First Affiliated Hospital of USTC(University of Science and Technology of China), Hefei, Anhui
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Fujian Provincial Hospital, Fuzhou, Fujian
  - Shenzhen Second People's Hospital, Shenzhen, Guangdong
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Eye& ENT Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Zhongshan Hospital,Fudan University, Shanghai, Shanghai Municipality